CLINICAL TRIAL: NCT02268903
Title: Diuretic Versus Placebo in Pulmonary Embolism With Right Ventricular Enlargement: a Double-blind Randomized Controlled Study
Brief Title: Diuretic Versus Placebo in Pulmonary Embolism
Acronym: DiPER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOM 130519
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Embolism With Right Ventricle Enlargement
Keywords: Pulmonary Embolism; Right Ventricle failure; Diuretics
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diuretics (Active Comparator)
  Interventions: Drug: Diuretics : Furosemide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diuretics : Furosemide — Furosemide 80mg in one single direct intra venous injection
  Arms: Diuretics
Drug: Placebo — Placebo in one single direct intra venous injection
  Arms: Placebo

SUMMARY:
Pulmonary Embolism (PE) is a frequent and severe disease with an annual incidence of about 75000 cases in France and a short-term mortality rate of about 10%. Death is usually related to an acute right ventricular (RV) failure due to the increase in right ventricular afterload. Treatment of PE with RV failure consists in fluid expansion and thrombolysis in case of shock. However several studies suggest that fluid expansion may worsen acute RV failure by increasing RV dilatation and ischemia and left ventricular compression by RV dilatation. Thus, current guidelines regarding PE treatment remain unclear about the use of fluid expansion. In a preliminary study published by our group, we showed that diuretic treatment in the setting of PE with RV dilatation is safe and is associated with an increase in urine output, a decrease in heart rate and an increase in SpO2 in normotensive patients with oliguria. This may be related to the decrease of ventricular interdependence and enhancement of both LV and RV function.

The main objective of the study is to evaluate the 24-hours clinical benefit of furosemide in patients referred for acute PE with RV dilatation compared to placebo. The combination of urine output and sPESI clinical parameters reflects hemodynamic status. It is relevant as it indicates the disappearance of pre-shock symptoms and is therefore associated with a lower event risk. Thus, it allows early discharge of the patients from the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years and over with

1. Symptomatic acute pulmonary embolism with first clinical symptoms within 15 days, and objectively confirmed by CT scan
2. RV dysfunction (≥1 criterion) confirmed by elevated BNP value or echocardiography or spiral computed tomography of the chest:

   * Echocardiography

     o Right/Left ventricular end diastolic diameter > 1(apical or subcostal 4-chamber view)
   * Computed tomography

     o Right/Left short-axis diameter ratio>0.9 (transverse plane)
   * Positive Nt-proBNP (>600) or BNP>200 pg/mL
3. One abnormal following PESI criteria

   * Heart Rate>110/min
   * Systolic blood pressure<100mmHg
   * Arterial oxyhemoglobin level<90% on room air or after 5 minutes of oxygen withdrawal.

Exclusion Criteria:

* Cardiogenic shock requiring thrombolysis
* Previous significant left ventricular insufficiency (LVEF<45%)
* Systolic blood pressure<90mmHg at admission
* Age ≤ 18 years
* Pregnancy
* No health insurance
* Patients deprived of liberty or under legal protection
* Creatinin clearance <30mL/min/m²
* hypersensibility to furosemide or its excipients
* functional renal insufficiency
* Hepatic encephalopathy
* Urinary tracks obstruction
* Hypovolemia or dehydration.
* Sever hypokalemia (K+ < 3mmol/L)
* Severe hyponatremia (Na+ < 125mmol/L)
* Ongoing hepatitis and hepatic insufficiency severe in patients with renal insufficiency or dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2015-04-13 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Primary end point will be a combined clinical criterion, to reach the primary endpoint, patients have to meet all the following criteria: - Urine output> 0.5ml/kg/h - Normalization of clinical parameters of simplified PESI score | 24 hours
  Normalization of clinical parameters of simplified PESI score :
  * Heart Rate<110/min
  * Systolic blood pressure≥100mmHg
  * Arterial oxyhemoglobin level>90% on room air or after 5 minutes of oxygen withdrawal.

SECONDARY OUTCOMES:
patients have to meet all the four following criteria: - Urine output> 0.5ml/kg/h over 24 hours - Normalization of clinical parameters of simplified PESI score - Urine output | 48 hours
  Normalization of clinical parameters of simplified PESI score :
  * Heart Rate<110/min
  * Systolic blood pressure≥100mmHg
  * Arterial oxyhemoglobin level>90% on room air or after 5 minutes of oxygen withdrawal.
- Composite criteria including death, need for catecholamine, cardiac arrest and mechanical ventilation during hospitalization and at 1 month from inclusion - NYHA score | In hospital and 1 month
o RV/LV ratio and decrease from baseline o Systolic pulmonary pressure and decrease from baseline o Tricuspid annular plane systolic expansion (TAPSE) at o Tricuspid annular plane systolic expansion (TAPSE) variation from baseline | 24 hours abd 1 month
  RV/LV ratio (diameters and surfaces)
- NT-proBNP or BNP decrease at 24hours - Creatinin and liver enzymes variations at 24hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc DUBOIS-RANDE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Wood KE. Major pulmonary embolism: review of a pathophysiologic approach to the golden hour of hemodynamically significant pulmonary embolism. Chest. 2002 Mar;121(3):877-905. doi: 10.1378/chest.121.3.877. PMID 11888976
- [Background] Lee FA. Hemodynamics of the right ventricle in normal and disease states. Cardiol Clin. 1992 Feb;10(1):59-67. PMID 1739960
- [Background] Torbicki A, Perrier A, Konstantinides S, Agnelli G, Galie N, Pruszczyk P, Bengel F, Brady AJ, Ferreira D, Janssens U, Klepetko W, Mayer E, Remy-Jardin M, Bassand JP; ESC Committee for Practice Guidelines (CPG). Guidelines on the diagnosis and management of acute pulmonary embolism: the Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). Eur Heart J. 2008 Sep;29(18):2276-315. doi: 10.1093/eurheartj/ehn310. Epub 2008 Aug 30. PMID 18757870
- [Background] Perlroth DJ, Sanders GD, Gould MK. Effectiveness and cost-effectiveness of thrombolysis in submassive pulmonary embolism. Arch Intern Med. 2007 Jan 8;167(1):74-80. doi: 10.1001/archinte.167.1.74. PMID 17210881
- [Background] Goldhaber SZ, Haire WD, Feldstein ML, Miller M, Toltzis R, Smith JL, Taveira da Silva AM, Come PC, Lee RT, Parker JA, et al. Alteplase versus heparin in acute pulmonary embolism: randomised trial assessing right-ventricular function and pulmonary perfusion. Lancet. 1993 Feb 27;341(8844):507-11. doi: 10.1016/0140-6736(93)90274-k. PMID 8094768
- [Derived] Lim P, Delmas C, Sanchez O, Meneveau N, Rosario R, Bouvaist H, Bernard A, Mansourati J, Couturaud F, Sebbane M, Coste P, Rohel G, Tardy B, Biendel C, Lairez O, Ivanes F, Gallet R, Dubois-Rande JL, Fard D, Chatelier G, Simon T, Paul M, Natella PA, Layese R, Bastuji-Garin S. Diuretic vs. placebo in intermediate-risk acute pulmonary embolism: a randomized clinical trial. Eur Heart J Acute Cardiovasc Care. 2022 Jan 12;11(1):2-9. doi: 10.1093/ehjacc/zuab082. PMID 34632490
- [Derived] Gallet R, Meyer G, Ternacle J, Biendel C, Brunet A, Meneveau N, Rosario R, Couturaud F, Sebbane M, Lamblin N, Bouvaist H, Coste P, Maitre B, Bastuji-Garin S, Dubois-Rande JL, Lim P. Diuretic versus placebo in normotensive acute pulmonary embolism with right ventricular enlargement and injury: a double-blind randomised placebo controlled study. Protocol of the DiPER study. BMJ Open. 2015 May 22;5(5):e007466. doi: 10.1136/bmjopen-2014-007466. PMID 26002690